CLINICAL TRIAL: NCT03066076
Title: Prospective Randomized Clinical Trial of Total Thyroidectomy (Tx) Versus Thionamides (Anti-Thyroid Drugs) in Patients With Moderate-to-Severe Graves' Ophthalmopathy - a 1-year Follow-up
Brief Title: Total Thyroidectomy Versus Thionamides in Patients With Moderate-to-Severe Graves' Ophthalmopathy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Philipp Riss, Professor, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1839/2015; 2015-003515-38 (EudraCT Number)
Record Dates: First submitted 2017-01-27; First posted 2017-02-28 (Actual); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Graves Disease; Graves Ophthalmopathy; Graves' Ophthalmopathy Worsened
MeSH Terms: conditions — Graves Disease; Graves Ophthalmopathy | interventions — Antithyroid Agents; Methimazole; Propylthiouracil

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Observer blinded analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Thyroidectomy (Active Comparator): Total thyroidectomy
  Interventions: Drug: Antithyroid Drug
- Antithyroid drug (Active Comparator): Thiamazol, Propylthiouracil
  Interventions: Procedure: Total thyroidectomy

INTERVENTIONS:
Drug: Antithyroid Drug — Antithyroid drug
  Other Names: Thiamazol; Propylthiouracil
  Arms: Thyroidectomy
Procedure: Total thyroidectomy — Operation
  Arms: Antithyroid drug

SUMMARY:
Introduction: Graves disease (GD) is characterized by thyrotoxicosis and goiter, arising through circulating autoantibodies that bind to and stimulate the thyroid hormone receptor (TSHR). Graves' ophthalmopathy (GO) is characterized by inflammation, expansion of the extraocular muscles and an increase in retroorbital fat. There are currently three forms of therapies offered: anti-thyroid drugs (ATD) (thionamides), radioactive iodine (RAI) and total thyroidectomy (Tx). There is currently no consensus on the treatment of Grave's disease and GO.

Objective: To examine the difference in the outcome of GO in patients with moderate-to-severe GO, who receive Tx versus further ATD after suffering their first relapse of GO or in which GO stays the same following the initial decrease in ATD therapy after 6 months.

Methods: This prospective randomized clinical trial with observer blinded analysis will analyze 60 patients with moderate-to-severe GO who receive Tx versus ATD without surgery. Main outcome variables include: muscle index measurements via ultrasound and thyroid antibody levels. Additional outcome variables include: CAScore/NOSPECS score, superonasal index measurements via ultrasound and quality of life score.

DETAILED DESCRIPTION:
Introduction: Graves disease (GD) is characterized by thyrotoxicosis and goiter, arising through circulating autoantibodies that bind to and stimulate the thyroid hormone receptor (TSHR). Graves' ophthalmopathy (GO) is characterized by inflammation, expansion of the extraocular muscles and an increase in retroorbital fat. There are currently three forms of therapies offered: anti-thyroid drugs (ATD) (thionamides), radioactive iodine (RAI) and total thyroidectomy (Tx). There is currently no consensus on the treatment of Grave's disease and GO.

Objective: To examine the difference in the outcome of GO in patients with moderate-to-severe GO, who receive Tx versus further ATD after suffering their first relapse of GO or in which GO stays the same following the initial decrease in ATD therapy after 6 months.

Methods: This prospective randomized clinical trial with observer blinded analysis will analyze 60 patients with moderate-to-severe GO who receive Tx versus ATD without surgery. Main outcome variables include: muscle index measurements via ultrasound and thyroid antibody levels. Additional outcome variables include: CAScore/NOSPECS score, superonasal index measurements via ultrasound and quality of life score.

ELIGIBILITY:
Inclusion Criteria:

1. GD and GO onset < 12 months
2. no previous GD treatment other than antithyroid drugs (ATD)
3. first relapse after decrease of antithyroid medication within 4-6 months
4. GO treatment with glucocorticoids based on the Kahaly scheme
5. patients under ATD with normal thyroid function or subclinical hyperthyroid function and moderate-to-severe GO
6. clinically active inflammation according to CAScore (>3/7)
7. informed consent

Exclusion Criteria:

1. GD and GO onset > 12 months
2. more than one relapse of GO longer than 6 months from diagnosis
3. previous GD treatment by RAI or surgery
4. SNI greater than 7.0
5. urgent orbital decompression surgery
6. loss of vision
7. loss of visual field
8. loss of color vision
9. patients not receiving glucocorticoids for GO
10. cytological findings of postsurgical histopathological results suspicious for malignancy
11. pregnancy or breast-feeding
12. contraindication to GC
13. halt of GC therapy
14. Patients with diabetes mellitus
15. age below 18 years
16. no informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-03-01 (Estimated); Primary Completion 2019-02-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Muscle index (MI) from ultrasound measurements | 12 months
  Muscle index (MI) from ultrasound measurements
Thyroid antibodies | 12 months
  Thyroid antibodies

SECONDARY OUTCOMES:
CAScore/NOSPECS score | 12 months
  CAScore/NOSPECS score
Superonasal index measurements via ultrasound | 12 months
  Superonasal index measurements via ultrasound
Quality of life score | 12 months
  Quality of life score

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Riss, MD, Principal Investigator — Medical University Vienna; Guido Dorner, MD, Principal Investigator — Medical University Vienna
Locations (1):
- Department of Surgery and Department of Ophthalmology Medical University Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
No IPD sharing